CLINICAL TRIAL: NCT02500927
Title: Phase II Study of ASP8273 - An Open-Label, Study of the Oral Administration of ASP8273 in Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor-NaïvePatients With Non-Small Cell Lung Cancer Harboring EGFR Mutations
Brief Title: A Study of ASP8273 in Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor-Naïve Patients With Non-Small Cell Lung Cancer Harboring EGFR Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies.
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0202
Record Dates: First submitted 2015-06-25; First posted 2015-07-17 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: EGFR-TKI-naïve Patients With NSCLC Harboring EGFR Activating Mutations
Keywords: ASP8273; Non-Small Cell Lung Cancer; EGFR Tyrosine Kinase Inhibitor; EGFR Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naquotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP8273 group (Experimental): Single oral administration of ASP8273 Capsule A for bioavailability evaluation, followed once daily multiple administration of ASP8273 Capsule
  Interventions: Drug: ASP8273 Capsules; Drug: ASP8273 Capsules A

INTERVENTIONS:
Drug: ASP8273 Capsules — oral
Drug: ASP8273 Capsules A — oral

SUMMARY:
The purpose of this study is to determine the safety, the antitumor activity and the pharmacokinetics of ASP8273 in EGFR tyrosine kinase inhibitor (EGFR-TKI)-naïve patients with non-small cell lung cancer (NSCLC) harboring EGFR activating mutations.

DETAILED DESCRIPTION:
This study consists of a single-dose period (Cycle 0 lasting 3 days) and a multiple-dose period (from Cycle 1 onwards, each cycle lasting 21 days). To compare the PK between ASP8273 Capsules and ASP8273 Capsules A, enrolled subjects will receive a single oral dose of ASP8273 Capsules A on Day 1 of Cycle 0 in the single-dose period and will then be observed for 3 days (including the day of dosing). In the multiple-dose period, subjects will receive multiple oral doses of ASP8273 Capsules during each cycle lasting 21 days. From the viewpoint of PK comparison (bioavailability [BA] evaluation) between ASP8273 Capsules and ASP8273 Capsules A, data from approximately 15 subjects are sufficient for the evaluation. Therefore, if PK data of approximately 15 subjects included in BA evaluation are obtained and the sponsor judges that further acquisition of PK data is not necessary, the single-dose period will not be conducted in subjects who are enrolled thereafter (subjects not included in BA evaluation). Subjects will continue to receive treatment with ASP8273 until they meet the discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Patients with a histologically or cytologically confirmed diagnosis of Stage IIIB or IV NSCLC.
* Patients confirmed to have the deletion of exon 19 (del ex19), L858R, G719X, or L861Q mutation among the EGFR activating mutations (patients at the study site who are documented to have any of the above-stated EGFR activating mutations can be enrolled in the study).
* Patients with a life expectancy ≥ 12 weeks based on the principal investigator's/subinvestigator's judgment.
* Patients who meet all of the following requirements for laboratory tests within 7 days before enrollment. When 2 or more test results for a single parameter are found within the specified period, the last data before enrollment should be used for assessment.

  * Neutrophil count: ≥ 1,500/mm3
  * Platelet count: ≥ 75,000/mm3
  * Hemoglobin: ≥ 9 g/dL
  * Serum creatinine: < 1.5 mg/dL
  * Total bilirubin (TBL): < 1.5 × the upper limit of normal (ULN) at the site (this does not apply to patients with Gilbert syndrome)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): < 2.5 ×the ULN at the site
* Patients who meet all the following requirements for prior treatment for NSCLC:

  * Patients who have not received previous treatment with EGFR-TKIs*1 *1: Erlotinib, gefitinib, afatinib, and EGFR-TKIs under clinical investigation (e.g.,neratinib, dacomitinib). EGFR-TKIs that can inhibit EGFR with the T790Mmutation (e.g., ASP8273, CO-1686, AZD9291) are also included.
* Patients who have not received more than one regimen of previous drug treatment (however, this does not include preoperative or postoperative therapies used within at least a 6-month interval after the last dose of the treatment).
* Patients who have at least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

Exclusion Criteria:

* Patients with persistent clinical evidence of previous antitumor treatment-related toxicity ≥ Grade 2 using the Japan Clinical Oncology Group (JCOG) Japanese translation of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (NCI CTCAE v4.0 - JCOG) (except alopecia).
* Patients with a history of or concurrent interstitial lung disease.
* Patients who have received previous treatment with intended antitumor effects or treatment with another investigational drug/medical device within 14 days before the start of the study treatment.
* Patients who have received transfusion or hematopoietic growth factor therapy within 14 days prior to the start of the study treatment.
* Patients who have received oral or intravenous corticosteroids within 7 days prior to the start of the study treatment (except to treat or prevent an allergic reaction).
* Patients who are scheduled to undergo a surgical procedure during the course of the study or the patient still has an unhealed wound after previous surgery.
* Patients with a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV).
* Patients with a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Patients with symptomatic central nervous system (CNS) lesions.
* Patients with a known history of serious drug hypersensitivity.
* Patients with evidence of active infection requiring systemic drug therapy within 14 days prior to the start of the study treatment.
* Patients who have received strong CYP3A inhibitors within 9 days prior to the start of the study treatment (for itraconazole, within 14 days prior to the start of the study treatment).
* Patients who have received moderate CYP3A inhibitors within 9 days prior to the start of the study treatment (only for subjects included in BA evaluation).
* Patients who have received strong or moderate CYP3A inducers within 14 days prior to the start of the study treatment (only for subjects included in BA evaluation).
* Patients with prolongation of the QTc interval (male: ≥ 451 ms, female: ≥ 471 ms) on the 12-lead electrocardiogram (ECG) in the screening period.
* Patients with cardiac arrhythmias requiring treatment.
* Patients with Class 3 or 4 New York Heart Association (NYHA) congestive heart failure.
* Patients with a history of acute coronary syndrome, myocardial infarction, or cerebrovascular accident within 6 months prior to enrollment.
* Patients with a history of or concurrent active peptic ulcer disease or gastrointestinal bleeding within 3 months prior to enrollment.
* Patients with corneal disease ≥ Grade 2.
* Patients with difficulty to take oral medication, or any gastrointestinal malfunction or inflammatory bowel disease that is considered to affect drug absorption.
* Patients with active multiple cancers (simultaneous multiple cancers).
* Patients with other conditions ineligible for participation in the study based on the principal investigator's/sub-investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Safety assessed by AEs | Up to 18 months
Safety assessed by Laboratory tests | Up to 18 months
Safety assessed by Vital signs | Up to 18 months
Safety assessed by Percutaneous oxygen saturation (SpO2) | Up to 18 months
Safety assessed by Body weight | Up to 18 months
Safety assessed by 12-lead ECG | Up to 18 months
  ECG: Electrocardiogram
Safety assessed by Ophthalmologic examination | Up to 18 months
Safety assessed by Chest X-ray examination | Up to 18 months
Safety assessed by Chest computed tomography (CT) examination | Up to 18 months
Safety assessed by ECOG Performance Status | Up to 18 months

SECONDARY OUTCOMES:
Overall response rate | Up to 18 months
  The overall response rate is defined as the proportion of subjects whose best overall response is rated as Complete response (CR) or Partial Response (PR)among all analyzed subjects
Disease control rate | Up to 18 months
  The disease control rate is defined as the proportion of subjects whose best overall response is rated as Complete response (CR), Partial Response (PR), or Stable disease (SD) among all analyzed subjects
Plasma concentrations of unchanged ASP8273 | Up to Day1 of Cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (11):
- Japan (11):
  - Site: 5, Fukuoka
  - Site: 9, Hiroshima
  - Site: 8, Hyōgo
  - Site: 7, Kanagawa
  - Site: 11, Miyagi
  - Site: 1, Miyagi
  - Site: 10, Nagoya
  - Site: 4, Okayama
  - Site: 3, Osaka
  - Site: 6, Osaka
  - Site: 2, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Azuma K, Nishio M, Hayashi H, Kiura K, Satouchi M, Sugawara S, Hida T, Iwamoto Y, Inoue A, Takeda K, Ikeda S, Nakagawa T, Takeda K, Asahina S, Komatsu K, Morita S, Fukuoka M, Nakagawa K. ASP8273 tolerability and antitumor activity in tyrosine kinase inhibitor-naive Japanese patients with EGFR mutation-positive non-small-cell lung cancer. Cancer Sci. 2018 Aug;109(8):2532-2538. doi: 10.1111/cas.13651. Epub 2018 Jun 29. PMID 29807396
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=258